CLINICAL TRIAL: NCT04400617
Title: Understanding the Association Between Sleep Quality, Physical Activity, and Memory in Assisted-Living Residents
Brief Title: Sleep Quality in Assisted-Living Residents
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Collaborators: The Brenda Strafford Foundation (Unknown)
Responsible Party: Principal Investigator, Marc Poulin, Professor, University of Calgary
Other Study IDs: REB 19-1939
Record Dates: First submitted 2020-05-14; First posted 2020-05-22 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Sleep Disturbance; Aging
Keywords: Sleep; Functional Capacity; Cognitive Performance; Assisted-Living Facilities
MeSH Terms: conditions — Parasomnias | interventions — Functional Status

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Assisted-living residents: The target population will be inactive men and women residents of the Brenda Strafford Foundation (> 50 yrs. old). We expect the participants to be classified as inactivity, which will be defined as an engagement in < 3 sessions/week of 20 min or more of vigorous exercise. Participants should be able to move independently without the assistance of a wheelchair.
  Interventions: Behavioral: Cross-sectional assessments to examine the relationship among sleep quality, functional/physical capacity, and cognitive performance.
- Control group: Volunteers from the Brain in Motion II (BIM II) study (NCT03035851). The BIM II study aims to examine the mechanisms whereby exercise may improve sleep and cognition in men and women aged 50 to 80 years old. As the baseline measurements of the BIM II study are similar to the assessments proposed in this study, the assisted living residents will be matched with older individuals of the same age and cognitive performance who live independently to answer the last research question.
  Interventions: Behavioral: Cross-sectional assessments to examine the relationship among sleep quality, functional/physical capacity, and cognitive performance.

INTERVENTIONS:
Behavioral: Cross-sectional assessments to examine the relationship among sleep quality, functional/physical capacity, and cognitive performance. — The first visit will consist of screening measurements. Participants will be asked to complete the following questionnaires: InterRAI Self Report Quality of Life Survey for Long Term Care Facilities (interRAI SQoL), Resident Assessment Instrument (RAI)-MDS 2.0, Global Physical Activity Questionnaire (GPAQ), Memory Complaint Questionnaire (MAC-Q), and Pittsburgh Sleep Quality Index (PSQI). At the end of this visit, the participants will be asked to wear the ActiWatch-2 (AW-2) as a wristwatch for 14 days. In the second visit, participants' height and weight will be measured and the participants will perform the following cognitive and functional tests: MoCA, Brief Visuospatial Memory Test-Revised (BVMT-R), Hopkins Verbal Learning Test-Revised (HVLT-R), Time up and Go (TUG), and Cognitive TUG (TUGcog). Finally, visit 3 will consist of on-site PSG recordings.

SUMMARY:
Assisted living residents who have sleep disturbances are at great risk of developing cognitive impairments. The identification of factors that increase sleep problems in this population is the first step towards improving sleep disorders and reducing and/or delaying the occurrence of cognitive impairments in this population. Physical activity has been proposed to improve sleep quality in older individuals, but there is currently no scientific evidence of how sleep mediates the relationship between physical activity and cognition in assisted living residents. This is a cross-sectional study that investigates the relationship between sleep quality, functional/physical capacity, and cognitive performance. Participants will be recruited through a non-probabilistic sampling method (convenience) as this is a feasibility study that aims to identify, for the first time, sleep disorders in assisted living residents using objective measures of sleep. Sleep quality will be measured with polysomnography, actigraphy, and questionnaire. Functional and physical capacity will be assessed through walking tasks and actigraphy. Cognitive tasks will be used to assess memory. This study will bring new insights into the factors that affect the quality of life and sleep in assisted living residents. The evidence-based knowledge acquired on-site will be translated and shared with the local and global scientific community to raise awareness of the factors that contribute to increasing institutionalization and dependent living. Results obtained from objective and subjective measures of sleep will be of great importance to develop specialized clinical expertise and behavioral interventions that will meet residents' needs.

DETAILED DESCRIPTION:
Specific Objectives and Hypotheses:

1. To test the feasibility of using polysomnography to identify the severity of sleep disorders in assisted living residents.

   The implementation of objective measures of sleep in assisted living residents is practical and provides accurate information on sleep architecture parameters.
2. To investigate the association between functional capacity and physical activity and sleep quality in assisted living residents using functional tests and actigraphy, respectively.

   There is a positive association between functional capacity and sleep quality and physical activity will improve sleep quality in the efficiency and duration domains.
3. To investigate the association between sleep quality, measured through actigraphy, and cognitive performance, specifically in the memory domain, in assisted living residents.

   There is a positive association between sleep quality, especially sleep efficiency, and cognitive performance.
4. To compare the sleep quality (measured with polysomnography, actigraphy, and questionnaire) in assisted living residents with older individuals of the same age and cognitive performance (Montreal Cognitive Assessment; MoCA score > 26) who live independently.

Sleep quality will be lower in assisted living residents in comparison with older individuals who live independently and the use of various methods to assess sleep quality will provide a better estimation of the differences in sleep quality between these populations.

ELIGIBILITY:
Inclusion Criteria:

* Be inactivity, which will be defined as an engagement in < 3 sessions/week of 20 min or more of vigorous exercise;
* Be able to move independently without the assistance of a wheelchair.

Exclusion Criteria:

* Diagnosis of a developmental handicap;
* Residents who are not able to understand communication and be understood by others and do not have decision-making capacity according to the Cognitive Performance Scale (CPS) > 3; The investigators will assess all the resident's capacity with the Brenda Strafford Foundation caregivers, even if their CPS is within the range included in the study (CPS 0-3);
* Terminal illness (life expectancy < 1 year);
* Not fluent in English;
* Currently participating in another trial;
* Comorbid medical or neurological illnesses (e.g., multiple sclerosis) that would confound cognitive assessments or make trial completion unlikely (in the site investigator's opinion);
* Contraindication for the tests.

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The target population will be inactive men and women residents of the Brenda Strafford Foundation (> 50 yrs. old).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Total sleep time. | Through study completion, an average of 1 year.
  The Prodigy Sleep Monitor (polysomnography) and Actiwatch 2 (actigraphy) will be used to analyze this sleep outcome.
Sleep efficiency. | Through study completion, an average of 1 year.
  The Prodigy Sleep Monitor (polysomnography) and Actiwatch 2 (actigraphy) will be used to analyze this sleep outcome.
Sleep onset latency. | Through study completion, an average of 1 year.
  The Prodigy Sleep Monitor (polysomnography) and Actiwatch 2 (actigraphy) will be used to analyze this sleep outcome.
Number of awakening. | Through study completion, an average of 1 year.
  The Prodigy Sleep Monitor (polysomnography) and Actiwatch 2 (actigraphy) will be used to analyze this sleep outcome.
PSQI component score. | Through study completion, an average of 1 year.
  The Pittsburgh Sleep Quality Index (PSQI) will be used to subjectively measure sleep quality and disturbances in the past few months. The self-related questions include the assessment of seven different sleep domains: sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction. The participant should score each of the seven areas from 0 (no difficulty) to 3 (severe difficulty). Final score ≥ 5 indicates poor sleep quality.

SECONDARY OUTCOMES:
Short-term memory, visuospatial ability, and executive function. | Through study completion, an average of 1 year.
  Montreal Cognitive Assessment (MoCA) will be used.
Visuo-spatial memory. | Through study completion, an average of 1 year.
  Visuospatial Memory Test-Revised (BVMT-R) will be used.
Verbal learning and memory. | Through study completion, an average of 1 year.
  Hopkins Verbal Learning Test-Revised (HVLT-R) will be used.
Functional capacity. | Through study completion, an average of 1 year.
  Time up and Go (TUG) task will be performed. The TUG test considers the time the participant takes to stand up from a chair, walk 3 m away, return to the chair, and sit down in the chair again.
Dual-task capacity. | Through study completion, an average of 1 year.
  Cognitive TUG (TUGcog) will be performed. In the TUGcog test, the participant should perform the same task while counting backward from a randomly assigned number between 60 and 100
Total number of counts (physical activity). | Through study completion, an average of 1 year.
  The Actiwatch 2 will be used for 14 days to record total movement and patterns of activity per day.

CONTACTS AND LOCATIONS:
Overall Officials: Marc J Poulin, PhD, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: No